CLINICAL TRIAL: NCT04642079
Title: A PHASE 3, SINGLE-ARM TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A 20-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN HEALTHY CHILDREN 15 MONTHS THROUGH 17 YEARS OF AGE
Brief Title: Safety and Immunogenicity Study of 20vPnC in Healthy Children 15 Months Through 17 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B7471014; 2019-003308-11 (EudraCT Number)
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Results first posted 2023-04-26 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: =>15 through 23 months of age (Experimental): 20vPnC
  Interventions: Biological: 20vPnC
- Cohort 2: 2 through 4 years of age (Experimental): 20vPnC
  Interventions: Biological: 20vPnC
- Cohort 3: 5 through 9 years of age (Experimental): 20vPnC
  Interventions: Biological: 20vPnC
- Cohort 4: 10 through 17 years of age (Experimental): 20vPnC
  Interventions: Biological: 20vPnC

INTERVENTIONS:
Biological: 20vPnC — 20-valent pneumococcal conjugate vaccine

SUMMARY:
This study is designed to evaluate the safety and immunogenicity of 20vPnC in healthy children 15 months through 17 years of age

ELIGIBILITY:
Inclusion Criteria:

* Male or female children ≥15 months to <18 years of age at the time of consent.
* Healthy children determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study.
* For children <5 years of age, written documentation of receipt of at least 3 doses of 13vPnC. The last dose of 13vPnC must have been administered >2 months before enrolment into the study

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis)
* Major known congenital malformation or serious chronic disorder
* Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results
* Previous vaccination with any investigational pneumococcal vaccine or with PPSV23, or planned receipt through study participation
* Cohorts 3 and 4: Pregnant or breastfeeding female participants

Ages: 15 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 839 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (42):
- United States (42):
  - Northwest Arkansas Pediatrics, Fayetteville, Arkansas
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - The Children's Clinic, Jonesboro, Arkansas
  - California Research Foundation, San Diego, California
  - Pharmax Research Clinic, Inc., Miami, Florida
  - Bio-Medical Research, LLC, Miami, Florida
  - Children's Health Center, Tampa, Florida
  - Tekton Research, Inc, Chamblee, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Meridian Clinical Research, LLC, Sioux City, Iowa
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - Michael W. Simon, M.D., PSC, Lexington, Kentucky
  - MedPharmics, LLC, Gulfport, Mississippi
  - Velocity Clinical Research, Grand Island, Grand Island, Nebraska
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Velocity Clinical Research, Norfolk, Norfolk, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Velocity Clinical Research, Sioux City, Omaha, Nebraska
  - Wr-Crcn, Llc, Henderson, Nevada
  - MedPharmic's, LLC, Albuquerque, New Mexico
  - Meridian Clinical Research, LLC, Binghamton, New York
  - Dayton Clinical Research, Dayton, Ohio
  - Ohio Pediatric Research Association Inc., Dayton, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - Allegheny Health and Wellness Pavilion, Erie, Pennsylvania
  - Lockman & Lubell Pediatric Associates, Fort Washington, Pennsylvania
  - Palmetto Pediatrics, PA, North Charleston, South Carolina
  - Benchmark Research, Austin, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Tekton Research, Inc, San Antonio, Texas
  - Alliance for Multispecialty Research, LLC, Layton, Utah
  - Wasatch Pediatrics, Cottonwood Office, Murray, Utah
  - Pediatric Care, Provo, Utah
  - JBR Clinical Research, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc./ Foothill Family Clinic South, Salt Lake City, Utah
  - CopperView Medical Center, South Jordan, Utah
  - J. Lewis Research, Inc. / Jordan River Family Medicine, South Jordan, Utah
  - Wee Care Pediatrics, Syracuse, Utah
  - Pediatric Associates of Charlottesville, PLC (Private Pediatric Practice), Charlottesville, Virginia
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471014

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 839 participants were enrolled and assigned to receive a single dose of 20-valent pneumococcal conjugate vaccine (20vPnC) of which 8 participants were not vaccinated and 831 were vaccinated with 20vPnC.
Groups:
- Cohort 1: 20vPnC: >=15 to <24 Months: Participants aged greater than or equal to (>=) 15 months to less than (<) 24 months who have been previously vaccinated with at least 3 doses of 13vPnC, were administered a single dose of 0.5 milliliter (mL) 20vPnC intramuscularly on Day 1. The last dose of 13vPnC must have been administered greater than (>) 2 months before enrollment into the study.
- Cohort 2: 20vPnC: >=2 to <5 Years: Participants aged >=2 to <5 years who have been previously vaccinated with at least 3 doses of 13vPnC, were administered a single dose of 0.5 mL 20vPnC intramuscularly on Day 1. The last dose of 13vPnC must have been administered >2 months before enrollment into the study.
- Cohort 3: 20vPnC: >=5 to <10 Years: Participants aged >=5 to <10 years regardless of previous vaccination status were administered a single dose of 0.5 mL 20vPnC intramuscularly on Day 1.
- Cohort 4: 20vPnC: >=10 to <18 Years: Participants aged >=10 to <18 years regardless of previous vaccination status were administered a single dose of 0.5 mL 20vPnC intramuscularly on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: 20vPnC: >=15 to <24 Months | Cohort 2: 20vPnC: >=2 to <5 Years | Cohort 3: 20vPnC: >=5 to <10 Years | Cohort 4: 20vPnC: >=10 to <18 Years
Started | 210 | 219 | 203 | 207
Vaccinated | 209 | 216 | 201 | 205
Completed | 207 | 210 | 199 | 203
Not Completed | 3 | 9 | 4 | 4
Not completed — Lost to Follow-up | 2 | 5 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 1 | 2
Not completed — Other | 0 | 0 | 0 | 1
Not completed — No longer met eligibility criteria | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Enrolled population included all participants who signed informed consent form (ICF).
Groups:
- Cohort 1: 20vPnC: >=15 to <24 Months: Participants aged greater than >=15 months to <24 months who have been previously vaccinated with at least 3 doses of 13vPnC, were administered a single dose of 0.5 mL 20vPnC intramuscularly on Day 1. The last dose of 13vPnC must have been administered >2 months before enrollment into the study.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 20vPnC: >=15 to <24 Months | Cohort 2: 20vPnC: >=2 to <5 Years | Cohort 3: 20vPnC: >=5 to <10 Years | Cohort 4: 20vPnC: >=10 to <18 Years | Total
Number analyzed (Participants) | 210 | 219 | 203 | 207 | 839
Age, Customized [Count of Participants; unit: Participants]
  28 Days to 23 Months | 210 | 0 | 0 | 0 | 210
  2 Years to 5 Years | 0 | 219 | 28 | 0 | 247
  6 Years to 11 Years | 0 | 0 | 175 | 51 | 226
  12 Years to 18 Years | 0 | 0 | 0 | 156 | 156
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 111 | 94 | 91 | 389
  Male | 117 | 108 | 109 | 116 | 450
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 46 | 32 | 45 | 158
  Not Hispanic or Latino | 173 | 173 | 169 | 161 | 676
  Unknown or Not Reported | 2 | 0 | 2 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 3 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 26 | 26 | 22 | 17 | 91
  White | 169 | 175 | 176 | 180 | 700
  More than one race | 10 | 14 | 5 | 9 | 38
  Unknown or Not Reported | 2 | 3 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Prompted Local Reactions Within 7 Days After Vaccination
Description: Local reactions included redness, swelling and, pain at the injection site, recorded by parent's/legal guardians of participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units. One measuring device unit =0.5 centimeter (cm). Redness and swelling were graded as mild: > 0.0 to 2.0 cm, moderate: >2.0 to 7.0 cm and severe: >7.0 cm. Pain at the injection site was graded as mild: hurt if gently touched (cohort 1) and did not interfere with activity (cohort 2-4); moderate: hurt if gently touched with crying (cohort 1) and interfered with daily activity (cohort 2-4) and; severe: limited limb movement (cohort 1) and prevented daily activity (cohort 2-4). 95 percent (%) confidence interval (CI) was based on Clopper and Pearson method.
Time Frame: Within 7 days after vaccination on Day 1
Population: Safety population included all participants who received 20vPnC and had safety follow-up after vaccination. Here, "Number of Participants Analyzed" signifies the number of participants with any electronic diary data after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: 20vPnC: >=15 to <24 Months | Cohort 2: 20vPnC: >=2 to <5 Years | Cohort 3: 20vPnC: >=5 to <10 Years | Cohort 4: 20vPnC: >=10 to <18 Years
Number analyzed (Participants) | 204 | 215 | 199 | 205
Percentage of participants
  Redness: Any | 37.7 [31.1 to 44.8] | 39.1 [32.5 to 45.9] | 37.2 [30.5 to 44.3] | 15.1 [10.5 to 20.8]
  Redness: Mild | 30.4 [24.2 to 37.2] | 22.8 [17.4 to 29.0] | 16.6 [11.7 to 22.5] | 10.7 [6.8 to 15.8]
  Redness: Moderate | 7.4 [4.2 to 11.8] | 15.3 [10.8 to 20.9] | 18.6 [13.4 to 24.7] | 3.9 [1.7 to 7.5]
  Redness: Severe | 0 [0.0 to 1.8] | 0.9 [0.1 to 3.3] | 2.0 [0.6 to 5.1] | 0.5 [0.0 to 2.7]
  Swelling: Any | 22.1 [16.6 to 28.4] | 23.3 [17.8 to 29.5] | 27.1 [21.1 to 33.9] | 15.6 [10.9 to 21.3]
  Swelling: Mild | 15.7 [11.0 to 21.4] | 11.6 [7.7 to 16.7] | 10.6 [6.7 to 15.7] | 5.4 [2.7 to 9.4]
  Swelling: Moderate | 6.4 [3.4 to 10.7] | 11.2 [7.3 to 16.2] | 15.6 [10.8 to 21.4] | 10.2 [6.5 to 15.2]
  Swelling: Severe | 0 [0.0 to 1.8] | 0.5 [0.0 to 2.6] | 1.0 [0.1 to 3.6] | 0 [0.0 to 1.8]
  Pain at the injection site: Any | 52.5 [45.4 to 59.5] | 66.0 [59.3 to 72.3] | 82.9 [77.0 to 87.9] | 82.0 [76.0 to 87.0]
  Pain at the injection site: Mild | 41.7 [34.8 to 48.8] | 47.0 [40.2 to 53.9] | 56.8 [49.6 to 63.8] | 62.9 [55.9 to 69.6]
  Pain at the injection site: Moderate | 9.8 [6.1 to 14.7] | 17.7 [12.8 to 23.4] | 24.6 [18.8 to 31.2] | 17.6 [12.6 to 23.5]
  Pain at the injection site: Severe | 1.0 [0.1 to 3.5] | 1.4 [0.3 to 4.0] | 1.5 [0.3 to 4.3] | 1.5 [0.3 to 4.2]

2. Primary Outcome: Percentage of Participants Reporting Prompted Systemic Events Within 7 Days After Vaccination: Cohort 1
Description: Systemic events for Cohort 1 included fever, decreased appetite, drowsiness/increased sleep and irritability, recorded by parents/legal guardians of participant's using an e-diary. Fever was defined as temperature >=38.0 degrees Celsius (C) and categorized as >=38.0 to 38.4 degrees C, >38.4 to 38.9 degrees C, >38.9 to 40.0 degrees C and >40.0-degrees C. Decreased appetite was graded as mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed). Drowsiness was graded as mild (increased or prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabling, not interested in usual daily activity). Irritability: graded as mild (easily consolable), moderate (required increased attention) and severe (inconsolable, crying could not be comforted). 95% CI was based on Clopper and Pearson method.
Time Frame: Within 7 days after vaccination on Day 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: 20vPnC: >=15 to <24 Months
Number analyzed (Participants) | 204
Percentage of participants
  Fever: >=38.0 degrees C | 11.8 [7.7 to 17.0]
  Fever: >=38.0 degrees C to 38.4 degrees C | 5.9 [3.1 to 10.0]
  Fever: >38.4 degrees C to 38.9 degrees C | 2.9 [1.1 to 6.3]
  Fever: >38.9 degrees C to 40.0 degrees C | 2.9 [1.1 to 6.3]
  Fever: >40.0 degrees C | 0 [0.0 to 1.8]
  Decreased appetite: Any | 25.0 [19.2 to 31.5]
  Decreased appetite: Mild | 17.6 [12.7 to 23.6]
  Decreased appetite: Moderate | 6.4 [3.4 to 10.7]
  Decreased appetite: Severe | 1.0 [0.1 to 3.5]
  Drowsiness/increased sleep: Any | 41.7 [34.8 to 48.8]
  Drowsiness/increased sleep: Mild | 31.4 [25.1 to 38.2]
  Drowsiness/increased sleep: Moderate | 9.3 [5.7 to 14.2]
  Drowsiness/increased sleep: Severe | 1.0 [0.1 to 3.5]
  Irritability: Any | 61.8 [54.7 to 68.5]
  Irritability: Mild | 22.5 [17.0 to 28.9]
  Irritability: Moderate | 37.3 [30.6 to 44.3]
  Irritability: Severe | 2.0 [0.5 to 4.9]

3. Primary Outcome: Percentage of Participants Reporting Prompted Systemic Events Within 7 Days After Vaccination: Cohorts 2, 3 and 4
Description: Systemic events for Cohort 2-4 included fever, fatigue, headache, muscle pain and joint pain, recorded by parents/legal guardians of participant's using an e-diary. Fever was defined as temperature >=38.0 degrees C and categorized as >=38.0 to 38.4 degrees C, >38.4 to 38.9 degrees C, >38.9 to 40.0 degrees C and >40.0 degrees C. Fatigue, headache, muscle pain and joint pain were graded as mild (no interference with activity), moderate (some interference with activity) and severe (prevents daily routine activity). 95% CI was based on Clopper and Pearson method.
Time Frame: Within 7 days after vaccination on Day 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: 20vPnC: >=2 to <5 Years | Cohort 3: 20vPnC: >=5 to <10 Years | Cohort 4: 20vPnC: >=10 to <18 Years
Number analyzed (Participants) | 215 | 199 | 205
Percentage of participants
  Fever: >=38.0 degrees C | 3.3 [1.3 to 6.6] | 0.5 [0.0 to 2.8] | 0 [0.0 to 1.8]
  Fever: >=38.0 degrees C to 38.4 degrees C | 1.4 [0.3 to 4.0] | 0.5 [0.0 to 2.8] | 0 [0.0 to 1.8]
  Fever: >38.4 degrees C to 38.9 degrees C | 1.4 [0.3 to 4.0] | 0 [0.0 to 1.8] | 0 [0.0 to 1.8]
  Fever: >38.9 degrees C to 40.0 degrees C | 0.5 [0.0 to 2.6] | 0 [0.0 to 1.8] | 0 [0.0 to 1.8]
  Fever: >40.0 degrees C | 0 [0.0 to 1.7] | 0 [0.0 to 1.8] | 0 [0.0 to 1.8]
  Fatigue: Any | 37.2 [30.7 to 44.0] | 28.1 [22.0 to 34.9] | 27.8 [21.8 to 34.5]
  Fatigue: Mild | 21.9 [16.5 to 28.0] | 19.1 [13.9 to 25.3] | 15.6 [10.9 to 21.3]
  Fatigue: Moderate | 14.4 [10.0 to 19.8] | 8.5 [5.1 to 13.3] | 12.2 [8.0 to 17.5]
  Fatigue: Severe | 0.9 [0.1 to 3.3] | 0.5 [0.0 to 2.8] | 0 [0.0 to 1.8]
  Headache: Any | 5.6 [2.9 to 9.5] | 18.6 [13.4 to 24.7] | 29.3 [23.1 to 36.0]
  Headache: Mild | 3.3 [1.3 to 6.6] | 14.6 [10.0 to 20.3] | 20.0 [14.8 to 26.1]
  Headache: Moderate | 1.9 [0.5 to 4.7] | 3.0 [1.1 to 6.4] | 7.8 [4.5 to 12.4]
  Headache: Severe | 0.5 [0.0 to 2.6] | 1.0 [0.1 to 3.6] | 1.5 [0.3 to 4.2]
  Muscle pain: Any | 26.5 [20.7 to 32.9] | 39.2 [32.4 to 46.3] | 48.3 [41.3 to 55.4]
  Muscle pain: Mild | 17.7 [12.8 to 23.4] | 26.6 [20.6 to 33.3] | 34.6 [28.1 to 41.6]
  Muscle pain: Moderate | 8.4 [5.0 to 12.9] | 11.1 [7.1 to 16.3] | 13.2 [8.9 to 18.6]
  Muscle pain: Severe | 0.5 [0.0 to 2.6] | 1.5 [0.3 to 4.3] | 0.5 [0.0 to 2.7]
  Joint pain: Any | 3.7 [1.6 to 7.2] | 6.5 [3.5 to 10.9] | 8.3 [4.9 to 12.9]
  Joint pain: Mild | 2.3 [0.8 to 5.3] | 3.0 [1.1 to 6.4] | 3.4 [1.4 to 6.9]
  Joint pain: Moderate | 1.4 [0.3 to 4.0] | 3.0 [1.1 to 6.4] | 4.9 [2.4 to 8.8]
  Joint pain: Severe | 0 [0.0 to 1.7] | 0.5 [0.0 to 2.8] | 0 [0.0 to 1.8]

4. Primary Outcome: Percentage of Participants Reporting Adverse Events (AEs) up to 1 Month After Vaccination
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. 95% CI was based on the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From vaccination (on Day 1) up to 1 month after vaccination
Population: Safety population included all participants who received 20vPnC and had safety follow-up after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: 20vPnC: >=15 to <24 Months | Cohort 2: 20vPnC: >=2 to <5 Years | Cohort 3: 20vPnC: >=5 to <10 Years | Cohort 4: 20vPnC: >=10 to <18 Years
Number analyzed (Participants) | 209 | 216 | 201 | 205
Percentage of participants | 23.9 (18.3) [18.3 to 30.3] | 7.9 (4.7) [4.7 to 12.3] | 6.5 (3.5) [3.5 to 10.8] | 4.4 (2.0) [2.0 to 8.2]

5. Primary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs) up to 6 Months After Vaccination
Description: An SAE was any untoward medical occurrence that occurred, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; was a congenital anomaly/birth defect and other important medical events. 95% CI was based on the Clopper and Pearson method.
Time Frame: From vaccination (on Day 1) up to 6 months after vaccination
Population: Safety population included all participants who received 20vPnC and had safety follow-up after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: 20vPnC: >=15 to <24 Months | Cohort 2: 20vPnC: >=2 to <5 Years | Cohort 3: 20vPnC: >=5 to <10 Years | Cohort 4: 20vPnC: >=10 to <18 Years
Number analyzed (Participants) | 209 | 216 | 201 | 205
Percentage of participants | 1.0 [0.1 to 3.4] | 0 [0.0 to 1.7] | 0 [0.0 to 1.8] | 1.5 [0.3 to 4.2]

6. Primary Outcome: Percentage of Participants Reporting Newly Diagnosed Chronic Medical Conditions (NDCMCs) up to 6 Months After Vaccination
Description: An NDCMC was defined as a disease or medical condition, not previously identified, that was expected to be persistent or was otherwise long-lasting in its effects. 95% CI was based on the Clopper and Pearson method.
Time Frame: From vaccination (on Day 1) up to 6 months after vaccination
Population: Safety population included all participants who received 20vPnC and had safety follow-up after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: 20vPnC: >=15 to <24 Months | Cohort 2: 20vPnC: >=2 to <5 Years | Cohort 3: 20vPnC: >=5 to <10 Years | Cohort 4: 20vPnC: >=10 to <18 Years
Number analyzed (Participants) | 209 | 216 | 201 | 205
Percentage of participants | 3.3 [1.4 to 6.8] | 0.5 [0.0 to 2.6] | 0.5 [0.0 to 2.7] | 1.0 [0.1 to 3.5]

7. Primary Outcome: Geometric Mean Fold Rises (GMFRs) of Pneumococcal Serotype-Specific Immunoglobulin G (IgG) Concentrations for the 7 Additional Serotypes From Before to 1 Month After 20vPnC Vaccination: Cohort 1 and 2
Description: Pneumococcal serotype-specific IgG concentrations were measured from serum samples for the 7 additional 20vPnC serotypes: 8, 10A, 11A, 12F, 15B, 22F and 33F. GMFR = geometric mean of fold rise from before vaccination on Day 1 to 1 month after vaccination with 20vPnC. GMFRs and corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of fold rises and the corresponding 2-sided 95% CIs (based on Student's t distribution). Superiority of IgG concentration 1 month after 20vPnC to before vaccination for each serotype was demonstrated if the 95% lower CI of GMFR was >1.
Time Frame: Before vaccination on Day 1 to 1 month after vaccination
Population: Evaluable immunogenicity population (EIP) included all participants who were eligible; received 20vPnC; at least 1 valid immunogenicity result from 1 month after vaccination collected within 27 to 56 days after vaccination for Cohorts 1-2; no other major protocol deviations. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants with valid assay results at both timepoints for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Cohort 1: 20vPnC: >=15 to <24 Months | Cohort 2: 20vPnC: >=2 to <5 Years
Number analyzed (Participants) | 188 | 182
Fold rise
  Serotype 8: number analyzed (Participants) | 186 | 178
  Serotype 8 | 113.4 [93.2 to 137.9] | 107.0 [86.1 to 133.0]
  Serotype 10A: number analyzed (Participants) | 188 | 181
  Serotype 10A | 83.2 [69.1 to 100.2] | 106.7 [86.2 to 132.0]
  Serotype 11A | 62.7 [49.9 to 78.8] | 43.6 [33.2 to 57.1]
  Serotype 12F | 27.9 [22.9 to 34.1] | 36.6 [30.1 to 44.7]
  Serotype 15B: number analyzed (Participants) | 188 | 180
  Serotype 15B | 52.1 [43.2 to 62.8] | 73.3 [58.7 to 91.5]
  Serotype 22F | 1847.7 [1481.3 to 2304.5] | 796.2 [577.1 to 1098.4]
  Serotype 33F | 113.5 [92.5 to 139.2] | 78.3 [61.6 to 99.5]

8. Primary Outcome: GMFRs of Pneumococcal Serotype-Specific Opsonophagocytic Activity (OPA) Titers for the 7 Additional Serotypes From Before to 1 Month After 20vPnC Vaccination: Cohort 3 and 4
Description: Pneumococcal serotype-specific OPA titers were measured from serum samples for 7 the additional 20vPnC serotypes: 8, 10A, 11A, 12F, 15B, 22F and 33F. GMFR = geometric mean of fold rise from before vaccination on Day 1 to 1 month after vaccination with 20vPnC. GMFRs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of fold rises and the corresponding 2-sided 95% CIs (based on the Student's t distribution). Superiority of OPA titers 1 month after 20vPnC to before vaccination for each serotype was demonstrated if the 95% lower CI of the GMFR was >1.
Time Frame: Before vaccination on Day 1 to 1 month after vaccination
Population: EIP included all participants who were eligible; received 20vPnC; at least 1 valid immunogenicity result from 1 month after vaccination collected within 27 to 49 days after vaccination for Cohorts 3-4; no other major protocol deviations. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants with valid assay results at both timepoints for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Cohort 3: 20vPnC: >=5 to <10 Years | Cohort 4: 20vPnC: >=10 to <18 Years
Number analyzed (Participants) | 154 | 174
Fold rise
  Serotype 8: number analyzed (Participants) | 153 | 174
  Serotype 8 | 106.5 [79.9 to 142.0] | 86.3 [64.2 to 115.9]
  Serotype 10A: number analyzed (Participants) | 134 | 142
  Serotype 10A | 30.6 [20.1 to 46.6] | 33.5 [22.3 to 50.1]
  Serotype 11A: number analyzed (Participants) | 136 | 155
  Serotype 11A | 11.6 [7.6 to 17.7] | 14.9 [10.2 to 21.8]
  Serotype 12F: number analyzed (Participants) | 154 | 164
  Serotype 12F | 463.6 [332.3 to 646.7] | 454.1 [333.3 to 618.7]
  Serotype 15B: number analyzed (Participants) | 142 | 164
  Serotype 15B | 380.8 [228.3 to 635.2] | 499.0 [338.7 to 735.3]
  Serotype 22F: number analyzed (Participants) | 137 | 168
  Serotype 22F | 128.5 [76.7 to 215.3] | 111.2 [67.1 to 184.3]
  Serotype 33F: number analyzed (Participants) | 144 | 158
  Serotype 33F | 14.2 [10.9 to 18.4] | 11.5 [8.9 to 14.9]

9. Secondary Outcome: Percentage of Participants With Predefined Levels of Pneumococcal Serotype-Specific IgG Concentrations for the 7 Additional Serotypes at 1 Month After Vaccination in Cohort 1 Only
Description: Pneumococcal serotype-specific IgG concentrations were measured from serum samples for the 7 additional 20vPnC serotypes: 8, 10A, 11A, 12F, 15B, 22F and 33F. Percentage of participants with predefined level (>=0.35 micrograms per milliliter) of IgG concentration for the 7 additional 20vPnC serotypes was presented. 2-sided 95% CI was based on Clopper and Pearson method.
Time Frame: At 1 Month after vaccination on Day 1
Population: EIP included all participants who were eligible; received 20vPnC; at least 1 valid immunogenicity result from 1 month after vaccination collected within 27 to 56 days after vaccination for Cohort 1; no other major protocol deviations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: 20vPnC: >=15 to <24 Months
Number analyzed (Participants) | 190
Percentage of participants
  Serotype 8 | 100.0 (98.1) [98.1 to 100.0]
  Serotype 10A | 83.2 (77.1) [77.1 to 88.2]
  Serotype 11A | 93.2 (88.6) [88.6 to 96.3]
  Serotype 12F | 40.0 (33.0) [33.0 to 47.3]
  Serotype 15B | 83.7 (77.6) [77.6 to 88.6]
  Serotype 22F | 98.9 (96.2) [96.2 to 99.9]
  Serotype 33F | 92.6 (87.9) [87.9 to 95.9]

10. Secondary Outcome: Percentage of Participants With >=4-fold Rise in Pneumococcal Serotype-Specific OPA Titers for the 7 Additional Serotypes From Before to 1 Month After Vaccination: Cohorts 2, 3, and 4 Only
Description: Pneumococcal serotype-specific OPA titers were measured from serum samples for 7 additional 20vPnC serotypes: 8, 10A, 11A, 12F, 15B, 22F and 33F. Percentage of participants with >=4-fold rise in serotype-specific OPA titers from before vaccination to 1 month after vaccination with 20vPnC and the associated 2-sided 95% CI based on the Clopper and Pearson method was presented. OPA titers were measured in a randomized subset of samples in Cohort 2 for this outcome measure.
Time Frame: Before vaccination on Day 1 to 1 month after vaccination
Population: EIP included all participants who were eligible; received 20vPnC;at least 1 valid immunogenicity result from 1 month after vaccination collected within 27 to 56 days or 27 to 49 days after vaccination for Cohort 2 or Cohorts 3-4, respectively; no other major protocol deviations. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants with valid assay results at both timepoints for the specified serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: 20vPnC: >=2 to <5 Years | Cohort 3: 20vPnC: >=5 to <10 Years | Cohort 4: 20vPnC: >=10 to <18 Years
Number analyzed (Participants) | 76 | 154 | 174
Percentage of participants
  Serotype 8: number analyzed (Participants) | 74 | 153 | 174
  Serotype 8 | 93.2 [84.9 to 97.8] | 92.2 [86.7 to 95.9] | 89.1 [83.5 to 93.3]
  Serotype 10A: number analyzed (Participants) | 73 | 134 | 142
  Serotype 10A | 84.9 [74.6 to 92.2] | 80.6 [72.9 to 86.9] | 81.7 [74.3 to 87.7]
  Serotype 11A: number analyzed (Participants) | 52 | 136 | 155
  Serotype 11A | 86.5 [74.2 to 94.4] | 66.2 [57.6 to 74.1] | 62.6 [54.5 to 70.2]
  Serotype: 12F: number analyzed (Participants) | 74 | 154 | 164
  Serotype: 12F | 94.6 [86.7 to 98.5] | 96.8 [92.6 to 98.9] | 94.5 [89.8 to 97.5]
  Serotype: 15B: number analyzed (Participants) | 76 | 142 | 164
  Serotype: 15B | 88.2 [78.7 to 94.4] | 89.4 [83.2 to 94.0] | 93.9 [89.1 to 97.0]
  Serotype: 22F: number analyzed (Participants) | 68 | 137 | 168
  Serotype: 22F | 86.8 [76.4 to 93.8] | 87.6 [80.9 to 92.6] | 81.0 [74.2 to 86.6]
  Serotype: 33F: number analyzed (Participants) | 73 | 144 | 158
  Serotype: 33F | 71.2 [59.4 to 81.2] | 79.9 [72.4 to 86.1] | 75.3 [67.8 to 81.8]

11. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Pneumococcal Serotype-Specific IgG for the 20vPnC Serotypes Before and 1 Month After Vaccination
Description: Pneumococcal serotype-specific IgG concentrations were measured for serum samples for 13vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F; and 7 additional 20vPnC serotypes: 8, 10A, 11A, 12F, 15B, 22F and 33F. GMCs the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding 2-sided 95% CIs (based on the Student's t distribution).
Time Frame: Before vaccination and 1 month after vaccination
Population: EIP included all participants who were eligible; received 20vPnC; at least 1 valid immunogenicity result from 1 month after vaccination collected within 27 to 56 days or within 27 to 49 days after vaccination for Cohorts 1-2 or Cohorts 3-4, respectively; no other major protocol deviations. Here, "Number of Participants Analyzed" signifies participants included in the EIP and "Number Analyzed" signifies participants with valid IgG concentrations at the specified timepoint for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter
Arm/Group | Cohort 1: 20vPnC: >=15 to <24 Months | Cohort 2: 20vPnC: >=2 to <5 Years | Cohort 3: 20vPnC: >=5 to <10 Years | Cohort 4: 20vPnC: >=10 to <18 Years
Number analyzed (Participants) | 190 | 183 | 186 | 198
Micrograms per milliliter
  Before Vaccination, Serotype 1: number analyzed (Participants) | 189 | 183 | 186 | 198
  Before Vaccination, Serotype 1 | 0.43 [0.37 to 0.49] | 0.20 [0.17 to 0.24] | 0.12 [0.10 to 0.14] | 0.09 [0.08 to 0.11]
  1 Month after Vaccination, Serotype 1 | 1.46 [1.28 to 1.67] | 4.21 [3.62 to 4.90] | 5.86 [5.15 to 6.67] | 4.04 [3.32 to 4.93]
  Before Vaccination, Serotype 3: number analyzed (Participants) | 189 | 183 | 186 | 198
  Before Vaccination, Serotype 3 | 0.14 [0.12 to 0.16] | 0.08 [0.06 to 0.10] | 0.22 [0.17 to 0.30] | 0.15 [0.11 to 0.20]
  1 Month after Vaccination, Serotype 3 | 0.54 [0.47 to 0.61] | 1.21 [1.04 to 1.42] | 1.32 [1.16 to 1.50] | 0.62 [0.52 to 0.76]
  Before Vaccination, Serotype 4: number analyzed (Participants) | 189 | 183 | 186 | 198
  Before Vaccination, Serotype 4 | 0.61 [0.52 to 0.72] | 0.30 [0.25 to 0.37] | 0.13 [0.11 to 0.16] | 0.12 [0.10 to 0.15]
  1 Month after Vaccination, Serotype 4 | 2.59 [2.27 to 2.96] | 8.37 [7.28 to 9.62] | 9.76 [8.54 to 11.15] | 6.37 [5.39 to 7.53]
  Before Vaccination, Serotype 5: number analyzed (Participants) | 189 | 183 | 186 | 198
  Before Vaccination, Serotype 5 | 0.43 [0.36 to 0.50] | 0.18 [0.15 to 0.22] | 0.07 [0.06 to 0.08] | 0.04 [0.03 to 0.06]
  1 Month after Vaccination, Serotype 5 | 1.53 [1.32 to 1.77] | 5.09 [4.32 to 5.99] | 7.50 [6.52 to 8.63] | 2.58 [1.88 to 3.53]
  Before Vaccination, Serotype 6A: number analyzed (Participants) | 188 | 183 | 184 | 195
  Before Vaccination, Serotype 6A | 1.61 [1.38 to 1.88] | 0.71 [0.58 to 0.88] | 0.50 [0.39 to 0.65] | 0.28 [0.22 to 0.37]
  1 Month after Vaccination, Serotype 6A | 7.59 [6.67 to 8.63] | 31.99 [27.85 to 36.75] | 46.28 [39.90 to 53.67] | 20.03 [15.39 to 26.07]
  Before Vaccination, Serotype 6B: number analyzed (Participants) | 188 | 183 | 182 | 195
  Before Vaccination, Serotype 6B | 0.85 [0.71 to 1.02] | 0.52 [0.42 to 0.63] | 0.26 [0.20 to 0.32] | 0.40 [0.31 to 0.51]
  1 Month after Vaccination, Serotype 6B | 4.27 [3.69 to 4.94] | 17.78 [15.43 to 20.48] | 32.45 [27.90 to 37.74] | 38.82 [31.49 to 47.86]
  Before Vaccination, Serotype 7F: number analyzed (Participants) | 189 | 183 | 186 | 198
  Before Vaccination, Serotype 7F | 1.17 [1.03 to 1.33] | 0.51 [0.44 to 0.60] | 0.18 [0.16 to 0.21] | 0.11 [0.08 to 0.14]
  1 Month after Vaccination, Serotype 7F | 3.53 [3.16 to 3.94] | 6.42 [5.69 to 7.24] | 7.92 [7.03 to 8.93] | 3.19 [2.65 to 3.85]
  Before Vaccination, Serotype 9V: number analyzed (Participants) | 189 | 183 | 186 | 198
  Before Vaccination, Serotype 9V | 0.71 [0.61 to 0.83] | 0.35 [0.28 to 0.42] | 0.14 [0.11 to 0.17] | 0.14 [0.11 to 0.18]
  1 Month after Vaccination, Serotype 9V | 2.70 [2.35 to 3.09] | 7.94 [6.83 to 9.24] | 10.86 [9.41 to 12.54] | 7.67 [6.52 to 9.02]
  Before Vaccination, Serotype 14: number analyzed (Participants) | 188 | 183 | 186 | 198
  Before Vaccination, Serotype 14 | 1.53 [1.31 to 1.79] | 0.66 [0.53 to 0.81] | 0.42 [0.33 to 0.53] | 0.29 [0.23 to 0.37]
  1 Month after Vaccination, Serotype 14: number analyzed (Participants) | 189 | 183 | 186 | 198
  1 Month after Vaccination, Serotype 14 | 4.42 [3.82 to 5.12] | 14.60 [12.44 to 17.13] | 28.54 [24.77 to 32.89] | 28.17 [23.90 to 33.21]
  Before Vaccination, Serotype 18C: number analyzed (Participants) | 189 | 183 | 186 | 198
  Before Vaccination, Serotype 18C | 0.65 [0.55 to 0.76] | 0.26 [0.21 to 0.32] | 0.12 [0.09 to 0.14] | 0.13 [0.11 to 0.17]
  1 Month after Vaccination, Serotype 18C | 2.69 [2.32 to 3.12] | 7.07 [6.01 to 8.32] | 10.83 [9.53 to 12.30] | 8.61 [7.34 to 10.10]
  Before Vaccination, Serotype 19A: number analyzed (Participants) | 189 | 183 | 186 | 198
  Before Vaccination, Serotype 19A | 0.47 [0.38 to 0.58] | 0.52 [0.40 to 0.68] | 0.78 [0.58 to 1.04] | 0.55 [0.43 to 0.70]
  1 Month after Vaccination, Serotype 19A: number analyzed (Participants) | 189 | 183 | 186 | 197
  1 Month after Vaccination, Serotype 19A | 3.29 [2.89 to 3.76] | 12.48 [10.76 to 14.48] | 13.65 [11.96 to 15.59] | 8.89 [7.29 to 10.84]
  Before Vaccination, Serotype 19F: number analyzed (Participants) | 189 | 183 | 186 | 198
  Before Vaccination, Serotype 19F | 0.80 [0.67 to 0.94] | 0.56 [0.44 to 0.71] | 0.96 [0.70 to 1.32] | 0.82 [0.63 to 1.06]
  1 Month after Vaccination, Serotype 19F | 4.16 [3.61 to 4.79] | 12.50 [10.48 to 14.91] | 14.62 [12.32 to 17.36] | 6.55 [5.60 to 7.66]
  Before Vaccination, Serotype 23F: number analyzed (Participants) | 189 | 183 | 186 | 198
  Before Vaccination, Serotype 23F | 0.96 [0.79 to 1.18] | 0.90 [0.71 to 1.15] | 0.82 [0.64 to 1.06] | 0.61 [0.48 to 0.78]
  1 Month after Vaccination, Serotype 23F | 5.35 [4.55 to 6.30] | 16.18 [13.75 to 19.04] | 22.69 [19.40 to 26.53] | 19.16 [16.31 to 22.51]
  Before Vaccination, Serotype 8: number analyzed (Participants) | 186 | 179 | 185 | 196
  Before Vaccination, Serotype 8 | 0.04 [0.03 to 0.05] | 0.05 [0.04 to 0.06] | 0.08 [0.07 to 0.10] | 0.16 [0.12 to 0.20]
  1 Month after Vaccination, Serotype 8: number analyzed (Participants) | 190 | 182 | 186 | 198
  1 Month after Vaccination, Serotype 8 | 4.66 [4.17 to 5.22] | 5.08 [4.45 to 5.80] | 4.65 [4.05 to 5.34] | 4.26 [3.67 to 4.94]
  Before Vaccination, Serotype 10A: number analyzed (Participants) | 188 | 183 | 186 | 198
  Before Vaccination, Serotype 10A | 0.01 [0.01 to 0.02] | 0.03 [0.02 to 0.03] | 0.07 [0.06 to 0.09] | 0.15 [0.12 to 0.19]
  1 Month after Vaccination, Serotype 10A: number analyzed (Participants) | 190 | 181 | 186 | 198
  1 Month after Vaccination, Serotype 10A | 1.23 [1.02 to 1.48] | 2.76 [2.28 to 3.34] | 3.98 [3.25 to 4.88] | 5.35 [4.20 to 6.81]
  Before Vaccination, Serotype 11A: number analyzed (Participants) | 188 | 183 | 186 | 198
  Before Vaccination, Serotype 11A | 0.03 [0.02 to 0.03] | 0.06 [0.04 to 0.08] | 0.12 [0.09 to 0.16] | 0.30 [0.23 to 0.38]
  1 Month after Vaccination, Serotype 11A: number analyzed (Participants) | 190 | 182 | 186 | 198
  1 Month after Vaccination, Serotype 11A | 1.61 [1.40 to 1.86] | 2.64 [2.25 to 3.09] | 2.80 [2.35 to 3.33] | 3.13 [2.60 to 3.77]
  Before Vaccination, Serotype 12F: number analyzed (Participants) | 188 | 183 | 186 | 198
  Before Vaccination, Serotype 12F | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01]
  1 Month after Vaccination, Serotype 12F: number analyzed (Participants) | 190 | 182 | 186 | 198
  1 Month after Vaccination, Serotype 12F | 0.22 [0.18 to 0.27] | 0.38 [0.31 to 0.46] | 0.36 [0.29 to 0.44] | 0.28 [0.22 to 0.34]
  Before Vaccination, Serotype 15B: number analyzed (Participants) | 188 | 182 | 186 | 198
  Before Vaccination, Serotype 15B | 0.02 [0.02 to 0.03] | 0.05 [0.04 to 0.07] | 0.20 [0.15 to 0.27] | 0.35 [0.27 to 0.45]
  1 Month after Vaccination, Serotype 15B: number analyzed (Participants) | 190 | 181 | 186 | 198
  1 Month after Vaccination, Serotype 15B | 1.17 [0.97 to 1.40] | 3.96 [3.12 to 5.03] | 10.74 [8.49 to 13.60] | 18.79 [15.16 to 23.28]
  Before Vaccination, Serotype 22F: number analyzed (Participants) | 188 | 183 | 186 | 198
  Before Vaccination, Serotype 22F | 0.01 [0.00 to 0.01] | 0.02 [0.01 to 0.02] | 0.08 [0.06 to 0.11] | 0.14 [0.11 to 0.19]
  1 Month after Vaccination, Serotype 22F: number analyzed (Participants) | 190 | 182 | 186 | 198
  1 Month after Vaccination, Serotype 22F | 9.57 [8.12 to 11.29] | 12.46 [10.82 to 14.35] | 15.68 [13.45 to 18.29] | 12.36 [10.38 to 14.72]
  Before Vaccination, Serotype 33F: number analyzed (Participants) | 188 | 183 | 185 | 196
  Before Vaccination, Serotype 33F | 0.02 [0.01 to 0.02] | 0.04 [0.03 to 0.05] | 0.10 [0.08 to 0.12] | 0.18 [0.14 to 0.22]
  1 Month after Vaccination, Serotype 33F: number analyzed (Participants) | 190 | 182 | 185 | 197
  1 Month after Vaccination, Serotype 33F | 1.91 [1.60 to 2.27] | 3.16 [2.63 to 3.79] | 3.87 [3.24 to 4.61] | 3.93 [3.25 to 4.75]

12. Secondary Outcome: GMFRs of Pneumococcal Serotype-Specific IgG Concentrations for the 13vPnC Serotypes From Before to 1 Month After Vaccination: Cohort 1 and 2
Description: Pneumococcal serotype-specific IgG concentrations were measured from serum samples for 13vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F. GMFR = geometric mean of fold rise from before vaccination on Day 1 to 1 month after vaccination with 20vPnC. GMFRs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the fold rises and the corresponding 2-sided 95% CIs (based on the Student's t distribution).
Time Frame: Before vaccination on Day 1 to 1 month after vaccination
Population: EIP included all participants who were eligible; received 20vPnC; at least 1 valid immunogenicity result from 1 month after vaccination collected within 27 to 56 days after vaccination for Cohorts 1-2; no other major protocol deviations. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants with valid assay results at both timepoints for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Cohort 1: 20vPnC: >=15 to <24 Months | Cohort 2: 20vPnC: >=2 to <5 Years
Number analyzed (Participants) | 189 | 183
Fold rise
  Serotype 1 | 3.4 [3.0 to 3.9] | 20.6 [17.2 to 24.7]
  Serotype 3 | 3.9 [3.4 to 4.5] | 14.9 [12.4 to 17.9]
  Serotype 4 | 4.3 [3.7 to 5.0] | 27.6 [22.7 to 33.5]
  Serotype 5 | 3.6 [3.1 to 4.2] | 28.2 [23.0 to 34.6]
  Serotype 6A: number analyzed (Participants) | 188 | 183
  Serotype 6A | 4.8 [4.1 to 5.6] | 44.9 [35.8 to 56.3]
  Serotype 6B: number analyzed (Participants) | 188 | 183
  Serotype 6B | 5.0 [4.3 to 5.9] | 34.5 [28.3 to 42.0]
  Serotype 7F | 3.0 [2.7 to 3.4] | 12.5 [10.5 to 14.9]
  Serotype 9V | 3.8 [3.3 to 4.4] | 23.0 [19.0 to 27.8]
  Serotype 14: number analyzed (Participants) | 187 | 183
  Serotype 14 | 2.9 [2.5 to 3.3] | 22.2 [18.0 to 27.4]
  Serotype 18C | 4.2 [3.6 to 4.9] | 27.2 [22.5 to 32.9]
  Serotype 19A: number analyzed (Participants) | 188 | 183
  Serotype 19A | 6.9 [5.7 to 8.4] | 24.1 [19.0 to 30.6]
  Serotype 19F | 5.2 [4.4 to 6.3] | 22.3 [17.2 to 28.8]
  Serotype 23F | 5.6 [4.8 to 6.6] | 17.9 [14.6 to 21.9]

13. Secondary Outcome: GMFRs of Pneumococcal Serotype-Specific IgG Concentrations for the 20vPnC Serotypes From Before to 1 Month After Vaccination: Cohort 3 and 4
Description: Pneumococcal serotype-specific IgG concentrations were measured from serum samples for 13vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F; and 7 additional 20vPnC serotypes: 8, 10A, 11A, 12F, 15B, 22F and 33F. GMFR = geometric mean of fold rise from before vaccination on Day 1 to 1 month after vaccination with 20vPnC. GMFRs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the fold rises and the corresponding 2-sided 95% CIs (based on the Student's t distribution).
Time Frame: Before vaccination on Day 1 to 1 month after vaccination
Population: EIP included all participants who were eligible; received 20vPnC; at least 1 valid immunogenicity result from 1 month after vaccination collected within 27 to 49 days after vaccination for Cohorts 3-4; no other major protocol deviations. Here, "Number of Participants Analyzed" signifies participants included in the EIP and "Number Analyzed" signifies participants with valid assay results at both timepoints for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Cohort 3: 20vPnC: >=5 to <10 Years | Cohort 4: 20vPnC: >=10 to <18 Years
Number analyzed (Participants) | 186 | 198
Fold rise
  Serotype 1 | 49.4 [41.6 to 58.6] | 44.2 [37.0 to 52.9]
  Serotype 3 | 5.9 [4.6 to 7.5] | 4.3 [3.5 to 5.2]
  Serotype 4 | 74.1 [61.4 to 89.4] | 52.0 [42.3 to 64.0]
  Serotype 5 | 107.0 [89.4 to 128.2] | 59.3 [47.6 to 73.9]
  Serotype 6A: number analyzed (Participants) | 184 | 195
  Serotype 6A | 91.9 [67.7 to 124.9] | 72.5 [54.9 to 95.7]
  Serotype 6B: number analyzed (Participants) | 182 | 195
  Serotype 6B | 127.9 [101.0 to 162.0] | 99.5 [77.1 to 128.3]
  Serotype 7F | 42.9 [36.1 to 51.1] | 30.0 [24.0 to 37.6]
  Serotype 9V | 80.3 [64.3 to 100.3] | 54.2 [42.7 to 68.9]
  Serotype 14 | 68.4 [53.4 to 87.7] | 96.7 [76.6 to 122.1]
  Serotype 18C | 93.7 [76.9 to 114.1] | 64.5 [52.3 to 79.4]
  Serotype 19A: number analyzed (Participants) | 186 | 197
  Serotype 19A | 17.6 [13.2 to 23.4] | 16.2 [13.1 to 20.0]
  Serotype 19F | 15.2 [10.5 to 22.0] | 8.0 [6.0 to 10.7]
  Serotype 23F | 27.6 [21.0 to 36.3] | 31.4 [23.8 to 41.5]
  Serotype 8: number analyzed (Participants) | 185 | 196
  Serotype 8 | 55.2 [44.8 to 67.9] | 27.3 [21.9 to 33.9]
  Serotype 10A | 54.8 [44.4 to 67.7] | 35.9 [29.3 to 43.9]
  Serotype 11A | 23.6 [18.6 to 29.9] | 10.5 [8.5 to 12.9]
  Serotype 12F | 31.9 [26.7 to 38.3] | 21.4 [17.6 to 26.0]
  Serotype 15B | 52.6 [41.3 to 66.9] | 53.8 [43.1 to 67.1]
  Serotype 22F | 187.7 [134.6 to 261.7] | 86.2 [64.9 to 114.4]
  Serotype 33F: number analyzed (Participants) | 184 | 195
  Serotype 33F | 39.3 [31.6 to 49.0] | 22.4 [18.2 to 27.6]

14. Secondary Outcome: Geometric Mean Titers (GMTs) of Pneumococcal Serotype-Specific OPA Titers for the 20vPnC Serotypes Before and 1 Month After Vaccination
Description: Pneumococcal serotype-specific OPA titers were measured from serum samples for 13vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F; and 7 additional 20vPnC serotypes: 8, 10A, 11A, 12F, 15B, 22F and 33F. GMTs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding 2-sided 95% CIs (based on the Student's t distribution). OPA titers were measured in a randomized subset of serum samples in Cohorts 1 and 2. OPA titers for the 13vPnC serotypes were measured in a randomized subset of serum samples in Cohorts 3 and 4.
Time Frame: Before vaccination on Day 1 and 1 month after vaccination
Population: EIP included all participants who were eligible; received 20vPnC; at least 1 valid immunogenicity result from 1 month after vaccination collected within 27 to 56 days or 27 to 49 days after vaccination for Cohorts 1-2 or Cohorts 3-4, respectively; no other major protocol deviations. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants with valid OPA titers at the specified timepoint for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: 20vPnC: >=15 to <24 Months | Cohort 2: 20vPnC: >=2 to <5 Years | Cohort 3: 20vPnC: >=5 to <10 Years | Cohort 4: 20vPnC: >=10 to <18 Years
Number analyzed (Participants) | 94 | 86 | 175 | 187
Titer
  Before Vaccination, Serotype 1: number analyzed (Participants) | 46 | 47 | 93 | 96
  Before Vaccination, Serotype 1 | 14 [11 to 18] | 12 [10 to 14] | 10 [9 to 11] | 11 [9 to 12]
  1 Month after Vaccination, Serotype 1: number analyzed (Participants) | 44 | 46 | 93 | 96
  1 Month after Vaccination, Serotype 1 | 57 [39 to 84] | 360 [272 to 476] | 548 [455 to 660] | 396 [302 to 519]
  Before Vaccination, Serotype 3: number analyzed (Participants) | 46 | 47 | 94 | 95
  Before Vaccination, Serotype 3 | 21 [15 to 29] | 15 [11 to 22] | 29 [22 to 40] | 19 [14 to 24]
  1 Month after Vaccination, Serotype 3: number analyzed (Participants) | 44 | 46 | 92 | 94
  1 Month after Vaccination, Serotype 3 | 80 [62 to 103] | 150 [116 to 195] | 155 [135 to 178] | 105 [88 to 124]
  Before Vaccination, Serotype 4: number analyzed (Participants) | 41 | 45 | 82 | 86
  Before Vaccination, Serotype 4 | 42 [24 to 75] | 34 [19 to 62] | 43 [27 to 67] | 34 [22 to 51]
  1 Month after Vaccination, Serotype 4: number analyzed (Participants) | 43 | 44 | 88 | 93
  1 Month after Vaccination, Serotype 4 | 563 [342 to 927] | 1729 [1188 to 2516] | 2328 [1942 to 2789] | 2290 [1822 to 2878]
  Before Vaccination, Serotype 5: number analyzed (Participants) | 46 | 47 | 94 | 96
  Before Vaccination, Serotype 5 | 18 [16 to 21] | 17 [15 to 20] | 15 [15 to 15] | 15 [15 to 16]
  1 Month after Vaccination, Serotype 5: number analyzed (Participants) | 44 | 46 | 92 | 96
  1 Month after Vaccination, Serotype 5 | 51 [38 to 68] | 198 [143 to 276] | 385 [324 to 458] | 216 [159 to 294]
  Before Vaccination, Serotype 6A: number analyzed (Participants) | 46 | 47 | 90 | 91
  Before Vaccination, Serotype 6A | 137 [77 to 243] | 96 [55 to 168] | 74 [51 to 106] | 64 [44 to 91]
  1 Month after Vaccination, Serotype 6A: number analyzed (Participants) | 43 | 46 | 92 | 96
  1 Month after Vaccination, Serotype 6A | 1707 [1144 to 2547] | 5283 [3954 to 7060] | 8268 [6617 to 10331] | 9434 [7616 to 11686]
  Before Vaccination, Serotype 6B: number analyzed (Participants) | 44 | 43 | 78 | 90
  Before Vaccination, Serotype 6B | 110 [67 to 182] | 126 [72 to 219] | 156 [99 to 244] | 237 [155 to 363]
  1 Month after Vaccination, Serotype 6B: number analyzed (Participants) | 44 | 46 | 90 | 93
  1 Month after Vaccination, Serotype 6B | 943 [611 to 1455] | 3273 [2390 to 4482] | 6569 [5367 to 8040] | 10085 [8263 to 12309]
  Before Vaccination, Serotype 7F: number analyzed (Participants) | 41 | 45 | 81 | 86
  Before Vaccination, Serotype 7F | 705 [492 to 1010] | 996 [748 to 1327] | 541 [410 to 713] | 516 [381 to 698]
  1 Month after Vaccination, Serotype 7F: number analyzed (Participants) | 42 | 44 | 87 | 93
  1 Month after Vaccination, Serotype 7F | 2635 [2105 to 3297] | 3409 [2552 to 4556] | 3981 [3446 to 4598] | 3326 [2878 to 3843]
  Before Vaccination, Serotype 9V: number analyzed (Participants) | 39 | 45 | 84 | 92
  Before Vaccination, Serotype 9V | 649 [350 to 1204] | 323 [202 to 515] | 410 [289 to 580] | 469 [330 to 667]
  1 Month after Vaccination, Serotype 9V: number analyzed (Participants) | 43 | 44 | 87 | 93
  1 Month after Vaccination, Serotype 9V | 7686 [5718 to 10332] | 7210 [4781 to 10876] | 11717 [9262 to 14823] | 9627 [7492 to 12369]
  Before Vaccination, Serotype 14: number analyzed (Participants) | 46 | 44 | 90 | 92
  Before Vaccination, Serotype 14 | 242 [151 to 387] | 300 [186 to 484] | 246 [172 to 353] | 97 [65 to 145]
  1 Month after Vaccination, Serotype 14: number analyzed (Participants) | 44 | 46 | 93 | 96
  1 Month after Vaccination, Serotype 14 | 1018 [748 to 1385] | 2506 [1932 to 3249] | 4610 [3688 to 5762] | 3925 [3153 to 4885]
  Before Vaccination, Serotype 18C: number analyzed (Participants) | 38 | 44 | 76 | 87
  Before Vaccination, Serotype 18C | 300 [147 to 613] | 139 [69 to 277] | 152 [89 to 261] | 73 [45 to 119]
  1 Month after Vaccination, Serotype 18C: number analyzed (Participants) | 43 | 44 | 87 | 93
  1 Month after Vaccination, Serotype 18C | 3749 [2740 to 5131] | 5344 [3809 to 7498] | 6766 [5585 to 8197] | 3617 [2816 to 4645]
  Before Vaccination, Serotype 19A: number analyzed (Participants) | 40 | 47 | 86 | 90
  Before Vaccination, Serotype 19A | 138 [71 to 271] | 84 [45 to 156] | 117 [76 to 181] | 66 [44 to 100]
  1 Month after Vaccination, Serotype 19A: number analyzed (Participants) | 43 | 44 | 88 | 93
  1 Month after Vaccination, Serotype 19A | 1708 [1192 to 2448] | 2640 [1943 to 3587] | 2162 [1786 to 2618] | 2212 [1801 to 2717]
  Before Vaccination, Serotype 19F: number analyzed (Participants) | 45 | 47 | 94 | 93
  Before Vaccination, Serotype 19F | 44 [31 to 61] | 44 [31 to 61] | 91 [66 to 125] | 57 [44 to 73]
  1 Month after Vaccination, Serotype 19F: number analyzed (Participants) | 44 | 46 | 92 | 96
  1 Month after Vaccination, Serotype 19F | 267 [169 to 421] | 928 [618 to 1394] | 1095 [810 to 1479] | 551 [401 to 757]
  Before Vaccination, Serotype 23F: number analyzed (Participants) | 41 | 46 | 87 | 92
  Before Vaccination, Serotype 23F | 139 [67 to 288] | 206 [108 to 394] | 87 [53 to 145] | 46 [29 to 73]
  1 Month after Vaccination, Serotype 23F: number analyzed (Participants) | 43 | 44 | 88 | 93
  1 Month after Vaccination, Serotype 23F | 1936 [1385 to 2707] | 2493 [1757 to 3539] | 2213 [1751 to 2797] | 1842 [1391 to 2439]
  Before Vaccination, Serotype 8: number analyzed (Participants) | 86 | 82 | 164 | 185
  Before Vaccination, Serotype 8 | 30 [24 to 39] | 39 [29 to 54] | 34 [28 to 42] | 35 [28 to 43]
  1 Month after Vaccination, Serotype 8: number analyzed (Participants) | 85 | 80 | 175 | 187
  1 Month after Vaccination, Serotype 8 | 4758 [3763 to 6016] | 4428 [3467 to 5654] | 3870 [3302 to 4535] | 3125 [2680 to 3642]
  Before Vaccination, Serotype 10A: number analyzed (Participants) | 84 | 82 | 158 | 168
  Before Vaccination, Serotype 10A | 92 [60 to 141] | 275 [160 to 472] | 745 [519 to 1071] | 554 [395 to 777]
  1 Month after Vaccination, Serotype 10A: number analyzed (Participants) | 86 | 78 | 159 | 171
  1 Month after Vaccination, Serotype 10A | 10626 [7825 to 14429] | 14345 [10473 to 19649] | 21102 [17238 to 25833] | 17417 [14301 to 21214]
  Before Vaccination, Serotype 11A: number analyzed (Participants) | 68 | 60 | 147 | 165
  Before Vaccination, Serotype 11A | 88 [60 to 127] | 436 [237 to 800] | 1347 [962 to 1887] | 765 [543 to 1076]
  1 Month after Vaccination, Serotype 11A: number analyzed (Participants) | 84 | 78 | 172 | 186
  1 Month after Vaccination, Serotype 11A | 13350 [10540 to 16910] | 14093 [9904 to 20054] | 16882 [13650 to 20880] | 11677 [9751 to 13982]
  Before Vaccination, Serotype 12F: number analyzed (Participants) | 92 | 86 | 174 | 182
  Before Vaccination, Serotype 12F | 38 [29 to 50] | 37 [27 to 50] | 48 [38 to 60] | 46 [36 to 59]
  1 Month after Vaccination, Serotype 12F: number analyzed (Participants) | 84 | 76 | 164 | 180
  1 Month after Vaccination, Serotype 12F | 16924 [13400 to 21376] | 13257 [9463 to 18572] | 23860 [19002 to 29959] | 20250 [16861 to 24320]
  Before Vaccination, Serotype 15B: number analyzed (Participants) | 94 | 84 | 163 | 187
  Before Vaccination, Serotype 15B | 30 [21 to 45] | 111 [63 to 197] | 79 [54 to 115] | 45 [33 to 61]
  1 Month after Vaccination, Serotype 15B: number analyzed (Participants) | 86 | 80 | 163 | 174
  1 Month after Vaccination, Serotype 15B | 22951 [17380 to 30307] | 27095 [19557 to 37538] | 25729 [19647 to 33695] | 21496 [16697 to 27672]
  Before Vaccination, Serotype: 22F: number analyzed (Participants) | 87 | 80 | 161 | 184
  Before Vaccination, Serotype: 22F | 21 [13 to 33] | 104 [55 to 194] | 259 [170 to 394] | 243 [161 to 366]
  1 Month after Vaccination, Serotype 22F: number analyzed (Participants) | 81 | 74 | 158 | 179
  1 Month after Vaccination, Serotype 22F | 22464 [16840 to 29967] | 25573 [18096 to 36141] | 33615 [26198 to 43130] | 27922 [22622 to 34463]
  Before Vaccination, Serotype: 33F: number analyzed (Participants) | 91 | 85 | 170 | 177
  Before Vaccination, Serotype: 33F | 1154 [861 to 1548] | 2179 [1694 to 2804] | 3334 [2847 to 3905] | 2895 [2448 to 3424]
  1 Month after Vaccination, Serotype 33F: number analyzed (Participants) | 81 | 76 | 155 | 171
  1 Month after Vaccination, Serotype 33F | 23431 [17375 to 31598] | 28076 [19255 to 40938] | 45921 [36768 to 57353] | 32363 [26219 to 39946]

15. Secondary Outcome: GMFRs of Pneumococcal Serotype-Specific OPA Titers for the 20vPnC Serotypes From Before to 1 Month After Vaccination: Cohorts 1 and 2
Description: Pneumococcal serotype-specific OPA titers were measured from serum samples for 13vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F; and 7 additional 20vPnC serotypes: 8, 10A, 11A, 12F, 15B, 22F and 33F. GMFR = geometric mean of fold rise from before vaccination on Day 1 to 1 month after vaccination with 20vPnC. GMFRs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the fold rises and the corresponding 2-sided 95% CIs (based on the Student's t distribution). OPA titers measured in a randomized subset of serum samples in Cohorts 1 and 2 for this outcome measure.
Time Frame: Before vaccination on Day 1 to 1 month after vaccination
Population: EIP included all participants who were eligible; received 20vPnC; at least 1 valid immunogenicity result from 1 month after vaccination collected within 27 to 56 days after vaccination for Cohorts 1-2; no other major protocol deviations. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants with valid assay results at both timepoints for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Cohort 1: 20vPnC: >=15 to <24 Months | Cohort 2: 20vPnC: >=2 to <5 Years
Number analyzed (Participants) | 84 | 76
Fold rise
  Serotype 1: number analyzed (Participants) | 42 | 46
  Serotype 1 | 4.1 [2.9 to 6.0] | 29.8 [21.2 to 41.9]
  Serotype 3: number analyzed (Participants) | 42 | 46
  Serotype 3 | 3.7 [2.6 to 5.3] | 9.6 [7.1 to 13.1]
  Serotype 4: number analyzed (Participants) | 40 | 41
  Serotype 4 | 13.2 [7.0 to 25.0] | 50.0 [26.7 to 93.6]
  Serotype 5: number analyzed (Participants) | 42 | 46
  Serotype 5 | 2.8 [2.0 to 3.8] | 11.4 [8.2 to 16.0]
  Serotype 6A: number analyzed (Participants) | 41 | 46
  Serotype 6A | 12.7 [8.1 to 20.0] | 52.9 [30.8 to 90.9]
  Serotype 6B: number analyzed (Participants) | 40 | 42
  Serotype 6B | 7.8 [4.6 to 13.2] | 24.4 [14.4 to 41.2]
  Serotype 7F: number analyzed (Participants) | 39 | 41
  Serotype 7F | 3.6 [2.5 to 5.2] | 3.6 [2.7 to 4.8]
  Serotype 9V: number analyzed (Participants) | 38 | 42
  Serotype 9V | 11.5 [6.2 to 21.3] | 23.1 [14.7 to 36.5]
  Serotype 14: number analyzed (Participants) | 42 | 43
  Serotype 14 | 3.9 [2.5 to 6.1] | 8.3 [5.1 to 13.4]
  Serotype 18C: number analyzed (Participants) | 38 | 40
  Serotype 18C | 12.7 [6.6 to 24.5] | 40.6 [20.7 to 79.6]
  Serotype 19A: number analyzed (Participants) | 39 | 43
  Serotype 19A | 11.1 [6.2 to 19.8] | 33.5 [17.3 to 65.0]
  Serotype 19F: number analyzed (Participants) | 41 | 46
  Serotype 19F | 5.7 [3.3 to 9.7] | 21.0 [13.0 to 33.9]
  Serotype 23F: number analyzed (Participants) | 40 | 42
  Serotype 23F | 12.5 [6.7 to 23.6] | 10.7 [6.2 to 18.5]
  Serotype 8: number analyzed (Participants) | 76 | 74
  Serotype 8 | 155.9 [110.4 to 220.2] | 105.4 [67.6 to 164.3]
  Serotype 10A: number analyzed (Participants) | 76 | 73
  Serotype 10A | 121.7 [74.7 to 198.4] | 53.3 [28.7 to 99.0]
  Serotype 11A: number analyzed (Participants) | 60 | 52
  Serotype 11A | 161.4 [115.7 to 225.2] | 34.7 [17.1 to 70.4]
  Serotype 12F: number analyzed (Participants) | 81 | 74
  Serotype 12F | 437.2 [307.0 to 622.7] | 319.9 [193.9 to 527.9]
  Serotype 15B | 717.6 [449.8 to 1144.6] | 294.4 [149.1 to 581.3]
  Serotype 22F: number analyzed (Participants) | 74 | 68
  Serotype 22F | 983.6 [580.9 to 1665.5] | 224.6 [104.9 to 480.9]
  Serotype 33F: number analyzed (Participants) | 78 | 73
  Serotype 33F | 18.8 [13.1 to 27.2] | 12.4 [7.4 to 20.7]

16. Secondary Outcome: GMFRs of Pneumococcal Serotype-Specific OPA Titers for the 13vPnC Serotypes From Before to 1 Month After Vaccination: Cohorts 3 and 4
Description: Pneumococcal serotype-specific OPA titers were measured for 13vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F. GMFR = geometric mean of fold rise from before vaccination on Day 1 to 1 month after vaccination with 20vPnC. GMFRs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the fold rises and the corresponding 2-sided 95% CIs (based on the Student's t distribution). OPA titers for the 13vPnC serotypes were measured in a randomized subset of serum samples in Cohorts 3 and 4.
Time Frame: Before vaccination on Day 1 to 1 month after vaccination
Population: EIP included all participants who were eligible; received 20vPnC; at least 1 valid immunogenicity result from 1 month after vaccination collected within 27 to 49 days after vaccination for Cohorts 3-4; no other major protocol deviations. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and " Number Analyzed" signifies participants with valid assay results at both timepoints for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Cohort 3: 20vPnC: >=5 to <10 Years | Cohort 4: 20vPnC: >=10 to <18 Years
Number analyzed (Participants) | 91 | 96
Fold rise
  Serotype 1 | 55.2 [45.1 to 67.4] | 37.3 [28.7 to 48.6]
  Serotype 3: number analyzed (Participants) | 91 | 93
  Serotype 3 | 5.3 [3.9 to 7.2] | 5.8 [4.5 to 7.5]
  Serotype 4: number analyzed (Participants) | 80 | 86
  Serotype 4 | 50.2 [31.6 to 79.5] | 65.6 [41.4 to 103.7]
  Serotype 5 | 26.7 [22.4 to 31.8] | 14.4 [10.5 to 19.6]
  Serotype 6A: number analyzed (Participants) | 87 | 91
  Serotype 6A | 110.3 [68.7 to 177.1] | 147.9 [96.0 to 228.0]
  Serotype 6B: number analyzed (Participants) | 73 | 87
  Serotype 6B | 38.8 [22.7 to 66.3] | 42.0 [26.1 to 67.6]
  Serotype 7F: number analyzed (Participants) | 78 | 86
  Serotype 7F | 7.0 [5.3 to 9.3] | 6.2 [4.4 to 8.8]
  Serotype 9V: number analyzed (Participants) | 82 | 92
  Serotype 9V | 28.9 [19.7 to 42.5] | 20.4 [13.4 to 31.0]
  Serotype 14: number analyzed (Participants) | 88 | 92
  Serotype 14 | 18.1 [12.2 to 26.8] | 38.9 [25.1 to 60.3]
  Serotype 18C: number analyzed (Participants) | 74 | 87
  Serotype 18C | 46.2 [26.8 to 79.6] | 47.3 [28.7 to 78.0]
  Serotype 19A: number analyzed (Participants) | 84 | 90
  Serotype 19A | 17.5 [10.8 to 28.3] | 33.1 [20.7 to 53.1]
  Serotype 19F: number analyzed (Participants) | 91 | 93
  Serotype 19F | 11.7 [7.4 to 18.5] | 10.0 [6.7 to 15.0]
  Serotype 23F: number analyzed (Participants) | 85 | 92
  Serotype 23F | 26.9 [16.3 to 44.5] | 39.4 [23.7 to 65.7]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events (systematic assessment): within 7 days after vaccination; SAEs (non-systematic assessment): from Day 1 up to 6 months after vaccination and other AEs (non-systematic assessment): from Day1 up to 1 month after vaccination
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Safety population included all participants who received 20vPnC and had safety follow-up after vaccination.
Arm/Group | Cohort 1: 20vPnC: >=15 to <24 Months | Cohort 2: 20vPnC: >=2 to <5 Years | Cohort 3: 20vPnC: >=5 to <10 Years | Cohort 4: 20vPnC: >=10 to <18 Years
All-Cause Mortality (participants affected / at risk) | 0/209 | 0/216 | 0/201 | 0/205
Serious Adverse Events (participants affected / at risk) | 2/209 | 0/216 | 0/201 | 3/205
Other Adverse Events (participants affected / at risk) | 173/209 | 163/216 | 178/201 | 186/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 20vPnC: >=15 to <24 Months (N=209) | Cohort 2: 20vPnC: >=2 to <5 Years (N=216) | Cohort 3: 20vPnC: >=5 to <10 Years (N=201) | Cohort 4: 20vPnC: >=10 to <18 Years (N=205)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Near drowning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 20vPnC: >=15 to <24 Months (N=209) | Cohort 2: 20vPnC: >=2 to <5 Years (N=216) | Cohort 3: 20vPnC: >=5 to <10 Years (N=201) | Cohort 4: 20vPnC: >=10 to <18 Years (N=205)
Injection site erythema (REDNESS) (General disorders) | 77 (84) | 84 (86) | 74 (79) | 31 (32)
Injection site pain (PAIN) (General disorders) | 107 (115) | 142 (157) | 165 (178) | 168 (175)
Injection site swelling (SWELLING) (General disorders) | 45 (51) | 50 (54) | 54 (57) | 32 (34)
Pyrexia (FEVER) (General disorders) | 24 (25) | 7 (9) | 1 (1) | 0 (0)
Decreased appetite (DECREASED APPETITE) (Metabolism and nutrition disorders) | 51 (72) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (9) | 13 (14) | 17 (17)
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 0 (0) | 57 (63) | 78 (86) | 99 (108)
Headache (HEADACHE) (Nervous system disorders) | 0 (0) | 12 (13) | 37 (45) | 60 (75)
Hypersomnia (INCREASED SLEEP) (Nervous system disorders) | 85 (104) | 0 (0) | 0 (0) | 0 (0)
Irritability (IRRITABILITY) (Psychiatric disorders) | 126 (170) | 0 (0) | 0 (0) | 0 (0)
Fatigue (FATIGUE) (General disorders) | 0 (0) | 80 (98) | 56 (76) | 57 (66)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT04642079/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT04642079/SAP_001.pdf